CLINICAL TRIAL: NCT02739984
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Safety, Tolerability, and Efficacy of Evolocumab (AMG 145) on LDL-C in Subjects With Type 2 Diabetes Mellitus and Hypercholesterolemia/Mixed Dyslipidemia
Brief Title: Evaluation of Evolocumab (AMG 145) Efficacy in Diabetic Adults With Hypercholesterolemia/Mixed Dyslipidemia
Acronym: BANTING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20130287; 2015-004711-21 (EudraCT Number)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hypercholesterolemia; Mixed Dyslipidemia; Type 2 Diabetes
Keywords: diabetes; type 2 diabetes; high blood cholesterol; hypercholesterolemia; mixed dyslipidemia; high cholesterol; statin intolerant
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once every month (QM) for 12 weeks.
  Interventions: Drug: Placebo to Evolocumab
- Evolocumab (Experimental): Participants received 420 mg evolocumab subcutaneous injection once every month (QM) for 12 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection with an automated mini doser
  Other Names: Repatha; AMG 145
  Arms: Evolocumab
Drug: Placebo to Evolocumab — Administered by subcutaneous injection with an automated mini doser
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of 12 weeks of subcutaneous evolocumab taken monthly compared with subcutaneous placebo taken monthly on low density lipoprotein cholesterol (LDL-C) in adults with type 2 diabetes mellitus and high blood cholesterol on a maximally tolerated oral dose of statin of at least moderate-intensity.

DETAILED DESCRIPTION:
This study will enroll adults with type 2 diabetes mellitus and elevated LDL-C or non-high-density lipoprotein cholesterol (non-HDL-C) levels on a stable, maximally tolerated statin dose of at least moderate-intensity at signing of the informed consent; statin therapy must remain unchanged during screening and the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* Type 2 Diabetes Mellitus
* Hemoglobin A1c < 10%
* Stable diabetes therapy
* Must be on maximally tolerated dose of statin of at least moderate Intensity
* Fasting triglycerides ≤ 600 mg/dL
* Not at LDL-C or Non-HDL-C goal.

Exclusion Criteria:

* Moderate to severe renal dysfunction
* Uncontrolled hypertension
* Persistent active liver disease or hepatic dysfunction
* Has taken a cholesterylester transfer protein inhibitor in the last 12 months,
* Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft or stroke within 3 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (61):
- United States (42):
  - Research Site, Tuscumbia, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Lomita, California
  - Research Site, Los Angeles, California
  - Research Site, Roseville, California
  - Research Site, San Ramon, California
  - Research Site, Spring Valley, California
  - Research Site, Tarzana, California
  - Research Site, Walnut Creek, California
  - Research Site, Denver, Colorado
  - Research Site, Lakewood, Colorado
  - Research Site, Wilmington, Delaware
  - Research Site, Boca Raton, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fleming Island, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Dunwoody, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Auburn, Maine
  - Research Site, Scarborough, Maine
  - Research Site, Salisbury, Maryland
  - Research Site, Methuen, Massachusetts
  - Research Site, Bay City, Michigan
  - Research Site, Tupelo, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Shelby, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Suffolk, Virginia
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
- Canada (4):
  - Research Site, Vancouver, British Columbia
  - Research Site, Gatineau, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jérôme, Quebec
- Italy (2):
  - Research Site, Roma
  - Research Site, Verona
- Mexico (2):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Chihuahua City
- Poland (4):
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Spain (4):
  - Research Site, Almería, Andalusia
  - Research Site, Granada, Andalusia
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia

REFERENCES:
- [Derived] Rosenson RS, Lopez JAG, Monsalvo ML, Wu Y, Wang H, Marcovina SM. Quantification of LDL-Cholesterol Corrected for Molar Concentration of Lipoprotein(a). Cardiovasc Drugs Ther. 2024 Feb;38(1):191-197. doi: 10.1007/s10557-022-07407-y. Epub 2022 Nov 26. PMID 36435949
- [Derived] Rosenson RS, Daviglus ML, Handelsman Y, Pozzilli P, Bays H, Monsalvo ML, Elliott-Davey M, Somaratne R, Reaven P. Efficacy and safety of evolocumab in individuals with type 2 diabetes mellitus: primary results of the randomised controlled BANTING study. Diabetologia. 2019 Jun;62(6):948-958. doi: 10.1007/s00125-019-4856-7. Epub 2019 Apr 5. PMID 30953107
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 853 patients screened, a total of 424 participants were randomized at 58 centers in Belgium, Canada, Italy, Mexico, Poland, Spain and the United States from 17 May 2016 to 05 May 2017.
Pre-assignment Details: Participants received subcutaneous placebo during a 6-week screening period. Participants who completed the screening period and met final eligibility criteria were randomized in a 1:2 ratio to placebo or evolocumab. Randomization was stratified by low-density lipoprotein cholesterol (LDL-C) level (> or < 130 mg/dL).
Period: Overall Study
Arm/Group | Placebo | Evolocumab
Started | 143 | 281
Received Study Drug | 141 | 280
Completed | 138 | 279
Not Completed | 5 | 2
Not completed — Sponsor Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab | Total
Number analyzed (Participants) | 143 | 281 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.5) | 62.5 (8.5) | 62.5 (8.5)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 86 | 159 | 245
  65 - < 85 years | 57 | 122 | 179
  ≥ 85 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 121 | 186
  Male | 78 | 160 | 238
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 54 | 78
  Not Hispanic or Latino | 119 | 227 | 346
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 8 | 15
  Asian | 2 | 4 | 6
  Black (or African American) | 32 | 41 | 73
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  White | 102 | 223 | 325
  Multiple | 0 | 1 | 1
  Other | 0 | 2 | 2
Stratification Factor: Low-density Lipoprotein Cholesterol (LDL-C) Level [Count of Participants; unit: Participants]
  < 130 mg/dL | 108 | 213 | 321
  ≥ 130 mg/dL | 35 | 68 | 103
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
  mg/dL
    number analyzed (Participants) | 141 | 280 | 421
    (all) | 110.4 (33.0) | 108.6 (31.0) | 109.2 (31.6)
Non-High-density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
  mg/dL
    number analyzed (Participants) | 141 | 280 | 421
    (all) | 145.5 (33.9) | 144.6 (34.9) | 144.9 (34.5)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab) and with available baseline data.
  mg/dL
    number analyzed (Participants) | 138 | 272 | 410
    (all) | 98.1 (22.1) | 97.1 (23.3) | 97.5 (22.9)
Total Cholesterol Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
  mg/dL
    number analyzed (Participants) | 141 | 280 | 421
    (all) | 190.7 (35.0) | 188.2 (36.8) | 189.1 (36.2)
Lipoprotein(a) Concentration [Mean (Standard Deviation); unit: nmol/L] — Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab) and with available baseline data.
  nmol/L
    number analyzed (Participants) | 137 | 273 | 410
    (all) | 99.4 (122.8) | 88.0 (111.5) | 91.8 (115.4)
Triglycerides Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
  mg/dL
    number analyzed (Participants) | 141 | 280 | 421
    (all) | 177.3 (89.2) | 184.2 (102.2) | 181.9 (98.0)
High-density Lipoprotein Cholesterol (HDL-C) Concentraion [Mean (Standard Deviation); unit: mg/dL] — Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
  mg/dL
    number analyzed (Participants) | 141 | 280 | 421
    (all) | 45.2 (12.2) | 43.6 (12.9) | 44.2 (12.7)
Very Low-density Lipoprotein Cholesterol (VLDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab) and with available baseline data.
  mg/dL
    number analyzed (Participants) | 138 | 276 | 414
    (all) | 33.6 (14.3) | 34.8 (15.4) | 34.4 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | -0.84 (1.76) | -64.98 (1.31)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; Model includes treatment group, stratification factor (screening LDL-C level), scheduled visit and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -64.14, 95% CI 2-sided [-68.16 to -60.12], Standard Error of Mean 2.05 — Evolocumab - Placebo

2. Primary Outcome: Percent Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | -1.14 (1.92) | -54.28 (1.42)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -53.14, 95% CI 2-sided [-57.56 to -48.71], Standard Error of Mean 2.25 — Evolocumab - Placebo

3. Secondary Outcome: Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
mg/dL | -8.3 (2.2) | -75.5 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -67.2, 95% CI 2-sided [-72.1 to -62.2], Standard Error of Mean 2.5 — Evolocumab - Placebo

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
mg/dL | -8.6 (2.3) | -64.4 (1.7)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.8, 95% CI 2-sided [-61.0 to -50.5], Standard Error of Mean 2.7 — Evolocumab - Placebo

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | -0.05 (1.63) | -56.62 (1.21)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.56, 95% CI 2-sided [-60.28 to -52.85], Standard Error of Mean 1.89 — Evolocumab - Placebo

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | -0.60 (1.79) | -46.89 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -46.28, 95% CI 2-sided [-50.42 to -42.15], Standard Error of Mean 2.10 — Evolocumab - Placebo

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | 2.31 (1.58) | -50.17 (1.18)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -52.48, 95% CI 2-sided [-56.10 to -48.85], Standard Error of Mean 1.85 — Evolocumab - Placebo

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | 1.78 (1.73) | -40.34 (1.29)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -42.12, 95% CI 2-sided [-46.13 to -38.11], Standard Error of Mean 2.04 — Evolocumab - Placebo

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | -1.13 (1.24) | -42.19 (0.92)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -41.06, 95% CI 2-sided [-43.90 to -38.22], Standard Error of Mean 1.44 — Evolocumab - Placebo

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | -1.23 (1.36) | -34.97 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.74, 95% CI 2-sided [-36.87 to -30.60], Standard Error of Mean 1.59 — Evolocumab - Placebo

11. Secondary Outcome: Percentage of Participants With Mean LDL-C at Weeks 10 and 12 Less Than 70 mg/dL (1.8 mmol/L)
Time Frame: Weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percentage of participants | 14.8 [9.8 to 21.8] | 92.7 [89.0 to 95.2]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel Haenszel (CMH) test adjusted by the stratification factor (screening LDL-C level); Treatment Difference = 77.9, 95% CI 2-sided [70.0 to 83.5] — Evolocumab - Placebo

12. Secondary Outcome: Percentage of Participants With LDL-C at Week 12 Less Than 70 mg/dL (1.8 mmol/L)
Time Frame: Week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percentage of participants | 15.4 [10.2 to 22.6] | 84.5 [79.5 to 88.5]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel Haenszel (CMH) test adjusted by the stratification factor (screening LDL-C level); Treatment Difference = 69.1, 95% CI 2-sided [60.4 to 75.7] — Evolocumab - Placebo

13. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in Mean LDL-C at Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percentage of participants | 0.7 [0.1 to 4.1] | 84.2 [79.5 to 88.1]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel Haenszel (CMH) test adjusted by the stratification factor (screening LDL-C level); Treatment Difference = 83.5, 95% CI 2-sided [77.7 to 87.4] — Evolocumab - Placebo

14. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in LDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percentage of participants | 0.8 [0.1 to 4.2] | 65.5 [59.4 to 71.1]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel Haenszel (CMH) test adjusted by the stratification factor (screening LDL-C level); Treatment Difference = 64.7, 95% CI 2-sided [57.7 to 70.3] — Evolocumab - Placebo

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | 9.63 (3.29) | -30.87 (2.43)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.50, 95% CI 2-sided [-48.11 to -32.90], Standard Error of Mean 3.87 — Evolocumab - Placebo

16. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | 7.38 (3.06) | -25.18 (2.28)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.56, 95% CI 2-sided [-39.58 to -25.53], Standard Error of Mean 3.57 — Evolocumab - Placebo

17. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | 6.61 (2.94) | -12.64 (2.19)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -19.25, 95% CI 2-sided [-25.95 to -12.54], Standard Error of Mean 3.41 — Evolocumab - Placebo

18. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | 4.81 (3.41) | -8.90 (2.52)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -13.70, 95% CI 2-sided [-21.60 to -5.80], Standard Error of Mean 4.02 — Evolocumab - Placebo

19. Secondary Outcome: Percent Change From Baseline in HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | -2.57 (1.25) | 7.23 (0.93)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 9.80, 95% CI 2-sided [6.95 to 12.64], Standard Error of Mean 1.45 — Evolocumab - Placebo

20. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | -1.41 (1.38) | 5.96 (1.02)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.37, 95% CI 2-sided [4.19 to 10.56], Standard Error of Mean 1.62 — Evolocumab - Placebo

21. Secondary Outcome: Percent Change From Baseline in VLDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | 3.42 (2.57) | -13.64 (1.89)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -17.06, 95% CI 2-sided [-22.91 to -11.21], Standard Error of Mean 2.98 — Evolocumab - Placebo

22. Secondary Outcome: Percent Change From Baseline in VLDL-C at Week 12
Time Frame: Baseline and week 12
Population: Randomized participants who received at least 1 dose of the study drug (placebo or evolocumab).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 141 | 280
percent change | 3.02 (2.94) | -10.31 (2.15)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -13.33, 95% CI 2-sided [-20.09 to -6.56], Standard Error of Mean 3.44 — Evolocumab - Placebo

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (placebo or evolocumab) to week 12.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Evolocumab
All-Cause Mortality (participants affected / at risk) | 0/141 | 1/280
Serious Adverse Events (participants affected / at risk) | 2/141 | 14/280
Other Adverse Events (participants affected / at risk) | 19/141 | 37/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=141) | Evolocumab (N=280)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=141) | Evolocumab (N=280)
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Pharyngitis (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 6
Viral upper respiratory tract infection (Infections and infestations) | 4 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 6
Hypertension (Vascular disorders) | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT02739984/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT02739984/SAP_001.pdf